CLINICAL TRIAL: NCT05144035
Title: A Real World Study of the Effect of Early PEG-rhGH Therapy on Cognitive Development of SGA Infants
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiaoping Luo, Director of Pediatrics, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gensci-GH-21005
Record Dates: First submitted 2021-10-17; First posted 2021-12-03 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Small for Gestational Age Infant; Growth Hormone Treatment; Cognitive Developmental Disorder
Keywords: SGA; PEG-rhGH; Cognitive developmental
MeSH Terms: interventions — polyethylene glycol-recombinant human growth hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GH treatment group (Experimental): GH treatment group (n = 68): the subjects were given PEG-rhGH injection 0.2 mg / kg / week (initial dose), once a week, subcutaneously before going to bed for 104 weeks. Each follow-up, the researchers adjusted the dosage according to the IGF-1 results of the center and other individual conditions.
  Interventions: Drug: PEG-rhGH
- Control group (No Intervention): Control group (n = 68): no treatment, only follow-up examination and growth and development related evaluation, and the follow-up time was 104 weeks.

INTERVENTIONS:
Drug: PEG-rhGH — the subjects were given PEG-rhGH injection 0.2 mg / kg / week (initial dose), once a week, subcutaneously before going to bed for 104 weeks. Each follow-up, the researchers adjusted the dosage according to the IGF-1 results of the center and other individual conditions.
  Other Names: jintrolong
  Arms: GH treatment group

SUMMARY:
Cognitive impairment is independently related to low birth weight, low birth length and small head circumference. SGA children who have not experienced height and / or head circumference catch-up have the worst cognitive function. The serum IGF-1 level of short SGA children is significantly lower than that of catch-up SGA children. This may be due to the defect of GH-IGF-1 axis, resulting in some hGH / IGF-1 deficiency.

GH treatment can induce catch-up growth of head circumference, especially for those with small birth head circumference, growth hormone can help to improve IQ, behavior and self cognition of children with SGA.

Two years after birth is the most critical period for children's physical, neurological, cognitive and emotional development. This study evaluated the effect of growth hormone treatment on the improvement of cognitive function and growth and development of symmetrical SGA children who did not show catch-up growth from 6 months to 2 years old.

This is an innovative study. The minimum age of previous similar studies is 19 months. The starting age of this study is 6 months, and the results are to improve the cognitive development of SGA infants. This is the first of its kind. Although the safety of growth hormone in SGA infants younger than 2 years old has not been reported, it is based on a number of studies on the application of growth hormone in infants, such as PWS and GHD, It can be expected that there will be no short-term and long-term adverse reactions.

The study was conducted in 17 hospitals led by Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of science and technology

DETAILED DESCRIPTION:
Subjects: SGA children from 6 months to 2 years old who meet the enrollment conditions shall be informed of the enrollment by the researcher and the subject's guardian, and the subject's guardian shall decide to participate in the test drug group or the control group.

GH treatment group (n = 68): the subjects were given PEG-rhGH injection 0.2 mg / kg / week (initial dose), once a week, subcutaneously before going to bed for 104 weeks. Each follow-up, the researchers adjusted the dosage according to the IGF-1 results of the center and other individual conditions.

Control group (n = 68): no treatment, only follow-up examination and growth and development related evaluation, and the follow-up time was 104 Week.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent signed and dated by the subject's legal guardian;
2. The subjects met the clinical diagnosis of small for gestational age infants.
3. The age ranged from 6 months to 2 years old (including 6 months and 2 years old);
4. Height and head circumference are lower than the reference value - 2sd (including-2sd), whose weight is lower than the 10th percentile of the reference value of normal children of the same age and sex;
5. The total developmental quotient GQ calculated according to Griffiths mental development scale is less than 100 points (100 points) Indicates that the developmental age is consistent with the physiological age);
6. Birth gestational age ≥ 37 weeks and < 42 weeks, single birth and non test tube baby;
7. Symmetrical SGA: birth weight index > 2.0 (gestational age = 37 weeks), or > 2.2 (gestational age > 37 weeks) . Weight index [birth weight (g) × 100 / birth length (CM) ];
8. Normal thyroid function or normal after replacement therapy;
9. No previous rhGH treatment

Exclusion Criteria:

1. Patients with abnormal liver and kidney function (ALT > 2 times the upper limit of normal value, Cr > the upper limit of normal value);
2. Severe familial dwarfism (father height < 155cm or mother height < 145cm);
3. Definite neurological defects and / or severe neurodevelopmental retardation (the total development quotient calculated according to Griffiths mental development scale is less than 70), definite syndrome affecting cognitive development; Severe perinatal complications (such as severe asphyxia, sepsis, necrotizing enterocolitis, respiratory distress syndrome with long-term sequelae);
4. Genetic metabolic diseases (such as congenital hypothyroidism, phenylketonuria, methylmalonic acidemia);
5. Congenital skeletal dysplasia, or moderate or above scoliosis (or scoliosis ≥ 15 °) requiring treatment or claudication;
6. Short stature with other definite causes, such as osteochondral dysplasia and Turner syndrome (TS), Noonan syndrome (NS), Prader Willi syndrome (PWS), Angelman syndrome (as), silver Russell syndrome (SRS), or other genetically confirmed syndromes (Note: diseases that meet the clinical diagnostic criteria adopt the method of clinical diagnosis; when the clinical diagnosis is difficult to be clear, or the diagnosis of the disease depends on gene screening, the method of gene diagnosis shall be supplemented / adopted);
7. patients with diabetes or fasting blood glucose are abnormal and the researchers believe that they may affect the safety of subjects.
8. Continuous application of other hormone therapy or systemic glucocorticoid therapy for more than one month in the past 6 months (local or inhaled glucocorticoids are allowed);
9. Patients with a history of convulsions or epilepsy, except for the relief or recovery of convulsions or epilepsy symptoms after the release of definite causes (such as high fever, calcium deficiency, brain infection, etc.);
10. Patients with other systemic chronic diseases;
11. Patients with confirmed tumors, or patients with family history of tumors (two or more tumor patients within three generations of immediate relatives), previous tumor history or considered as patients with high risk of tumors in combination with other information, clear syndromes with high risk of tumors (such as Bloom syndrome, Fanconi syndrome, Down syndrome, etc.);
12. Known high allergic constitution or allergic to the test drug in this study;
13. Those who have participated in clinical trials of other drugs within 3 months (the placebo group is not subject to this restriction);
14. Have received drug treatment that may interfere with GH secretion or GH effect within 3 months (including but not limited to any type of recombinant human growth hormone and protein assimilation drugs (including but not limited to oxandron, danazol and stanazol) other than rhGH injection);
15. The investigator considers that it is not suitable to be selected for this clinical trial.

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
total development quotient (GQ) | 104 weeks
  The changes of total development quotient (GQ) of young SGA children were calculated according to Griffiths mental development scale before and after treatment.（The Griffiths Scales,The normal range is from the 16th percentile to the 84th percentile of children of the same age. 100 is the mean. The higher the score, the better）
head circumference SDS | 104 weeks
  Changes of head circumference SDS in young SGA children before and after treatment

SECONDARY OUTCOMES:
Motor domain development quotient | 104 weeks
  Changes of motor domain development quotient (AQ) calculated according to Griffiths mental development scale before and after treatment.（The Griffiths Scales,The normal range is from the 16th percentile to the 84th percentile of children of the same age. 100 is the mean. The higher the score, the better）
Personal and social domain development quotient | 104 weeks
  Changes of personal and social domain development quotient (BQ) calculated according to Griffiths mental development scale before and after treatment.（The Griffiths Scales,The normal range is from the 16th percentile to the 84th percentile of children of the same age. 100 is the mean. The higher the score, the better）
Hearing and language domain development quotient | 104 weeks
  Changes of hearing and language domain development quotient (CQ) calculated according to Griffiths mental development scale before and after treatment.（The Griffiths Scales,The normal range is from the 16th percentile to the 84th percentile of children of the same age. 100 is the mean. The higher the score, the better）
Hand eye coordination domain development quotient | 104 weeks
  Changes of hand eye coordination domain development quotient (DQ) calculated according to Griffiths mental development scale before and after treatment.（The Griffiths Scales,The normal range is from the 16th percentile to the 84th percentile of children of the same age. 100 is the mean. The higher the score, the better）
Operation domain development quotient | 104 weeks
  Changes of operation domain development quotient (EQ) calculated according to Griffiths mental development scale before and after treatment.（The Griffiths Scales,The normal range is from the 16th percentile to the 84th percentile of children of the same age. 100 is the mean. The higher the score, the better）
Reasoning domain development quotient | 104 weeks
  Changes of reasoning domain development quotient (FQ) calculated according to Griffiths mental development scale before and after treatment.（The Griffiths Scales,The normal range is from the 16th percentile to the 84th percentile of children of the same age. 100 is the mean. The higher the score, the better）
Total T-scores and T-scores of behavior factors according to Achenbach children's behavior scale (CBCL).(The normal value is 100 points. The higher the score, the better) | 104 weeks
  Changes of total T-scores and T-scores of behavior factors calculated according to Achenbach children's behavior scale (CBCL) before and after treatment.(The normal value range is 55-70 points, and the lower the score, the better)
The adaptive behavior scale (ABAS-II) before and after treatment (GAC score) and three domain scores (cognitive skills, social skills and practical skills) | 104 weeks
  The adaptive comprehensive score was calculated according to the adaptive behavior scale (ABAS-II) before and after treatment.
  (The normal value is 100 points. The higher the score, the better)
height SDS | 104 weeks
  Changes of height SDS in young SGA children before and after treatment
Brain tissue metabolites | 104 weeks
  Brain tissue metabolites measured by cranial magnetic resonance spectroscopy (MRS) before and after treatment.
Myelin maturation | 104 weeks
  Myelin maturation was evaluated by diffusion tensor imaging (DTI) before and after treatment.
Brain volume and brain structure (Development) | 104 weeks
  Three dimensional T1 weighted imaging (3D) was performed before and after treatment T1WI) to assess brain volume and brain structure (Development).
Security | 104 weeks
  Related adverse reactions during the study

CONTACTS AND LOCATIONS:
Overall Officials: jianwei cao, director, Principal Investigator — Zhongshan People's Hospital (Zhongshan Hospital Affiliated to Sun Yat sen University)
Locations (1):
- Wuhan Tongji Hospital, Wuhan, Wuhan, China

IPD SHARING:
Plan to Share IPD: No